CLINICAL TRIAL: NCT05132998
Title: Impact of a Comprehensive Cardiac Rehabilitation Program Framework Among High Cardiovascular Risk Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associacao de Investigacao de Cuidados de Suporte em Oncologia (Other)
Collaborators: Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E. (Other Government); University Institute of Maia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CORE Trial
Record Dates: First submitted 2021-09-27; First posted 2021-11-24 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Oncologic Disorders; Cardiovascular Diseases
Keywords: cardiac rehabilitation; cardio-oncology rehabilitation; exercise training; cardiorespiratory fitness; cardiovascular risk factors
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac Rehabilitation Program (CRP) Group (Experimental): 1. Baseline consultation with physiatrist specialized in CRP - addressing CVRF control, comorbidities and disabilities; case-by-case discussion with a cardiologist specialized in CR will be undertaken, for tailoring exercise prescription. Nutritional individualized plan addressing dietary goals. Psychological management addressing psychosocial outcomes and motivation for healthy lifestyle habits
  2. Multidisciplinary team educational meeting: periodic group sessions with health education purposes
  3. Exercise intervention - 2 times/week sessions at CR facilities, supervised by a physiatrist, conducted by physiotherapist. Heart rate (HR) continuously monitored during each session by remote electrocardiographic monitoring or HR monitor. Exercise intensity estimated according to CR guidelines, determined after CV risk stratification, using CPET results.
  Interventions: Other: Cardiac Rehabilitation Program
- Community Exercise Group (Active Comparator): a) Besides standard medical and supportive care, psychological and nutritional individual support will be offered on demand, in hospital setting, according to the attending physician standard clinical assessment and usual care.
  Exercise intervention - Performed at a community-based facility, comprising 2 sessions/week, prescribed according to current physical activity guidelines for cancer survivors. Exercise intervention will be conducted by an exercise physiologist, internationally certified in exercise for cancer patients
  Interventions: Other: Community exercise intervention

INTERVENTIONS:
Other: Cardiac Rehabilitation Program — In addition to standard medical care, for an 8-week period, patients will have access to the core components of a CRP, delivered by a multidisciplinary rehabilitation team
  Arms: Cardiac Rehabilitation Program (CRP) Group
Other: Community exercise intervention — In addition to standard medical care, for an 8-week period, patients will have access to a community exercise intervention oriented by a sports professional
  Arms: Community Exercise Group

SUMMARY:
Many cancer survivors are at risk for cardiovascular disease (CVD); it is therefore important to identify patients at increased risk for cardiotoxicity, especially in the setting of CVRF or pre-existing CVD, and to design personalized interventions to prevent cardiovascular morbidity. In this background, cardio-oncology rehabilitation frameworks for specific cancer patients have been proposed. Given potential beneficial effects of exercise among cancer patients (including those at higher risk of CVD), data pertaining to optimal program designs are of paramount contemporary importance.

Thus, the aim of this study is to compare the impact of a Cardiac Rehabilitation Program (CRP) model versus a community-based exercise intervention plus usual care on cardiorespiratory fitness (CRF), physical function domains and CVRF control in adult cancer survivors who have been exposed to cardiotoxic cancer treatment and/or with cardiovascular medical background. Study outcomes will be assessed at baseline (M0) and after an 8 weeks-intervention (M1), comprising maximal aerobic capacity (peak oxygen uptake), muscular strength, neuromuscular function, single CVRF control including physical activity measurements and psychosocial parameters, health-related quality of life, fatigue, health literacy, inflammatory response and feasibility metrics; an economic evaluation will provide quantitative comparison, for a cost-effectiveness analysis

ELIGIBILITY:
Inclusion criteria:

* Age >18 years
* Cancer survivors exposed to the following therapies:

  * high-dose anthracycline or high dose radiotherapy in thoracic wall
  * low-dose anthracycline or anti-human Epidermal growth factor Receptor-type 2 drugs (anti-HER2) alone plus ≥ 2 CVRF and / or age ≥ 60 years at cancer treatment
  * low-dose anthracycline followed by anti-HER2;
* Cancer survivors with medical background of

  * coronary artery disease
  * moderate valvular disease
  * LVEF <50%
* Follow up after primary treatment with curative intent
* Conclusion of primary treatment at least 2 months before the inclusion

Exclusion criteria:

* Previous participation in a CRP
* Contraindications to exercise training:

  * musculoskeletal or neurologic disorders, cognitive impairment
  * unstable angor pectoris, decompensated HF, active myocarditis, acute endocarditis, acute pulmonary thromboembolism, complex ventricular arrhythmias
* Active cancer
* Considered unsuitable as per principal investigator judgment (namely due to expected inability to fulfill proposed schedule)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | Change from baseline to 2 months
  VO2peak measured by CPET

SECONDARY OUTCOMES:
Ventilatory efficiency | Change from baseline to 2 months
  minute ventilation to carbon dioxide production slope (VE/VCO2 slope) assessed by CPET
Sit-to-stand test | Change from baseline to 2 months
  Sit-to-stand test during 60 seconds
Handgrip maximal isometric muscle strength | Change from baseline to 2 months
  muscle strength measured with manual dynamometers (Kgf)
Body composition | Change from baseline to 2 months
  Changes in body composition assessed by bioelectrical impedance analysis
Resting diastolic blood pressure | Change from baseline to 2 months
  Measured with an average of 3 readings by an automated measurement device as per the ESC guidelines (mmHg)
Resting systolic blood pressure | Change from baseline to 2 months
  Measured with an average of 3 readings by an automated measurement device as per the ESC guidelines (mmHg)
Resting heart rate | Change from baseline to 2 months
  Measured with an average of 3 readings by an automated measurement device (bpm)
Hyperlipidemia | Change from baseline to 2 months
  Measured through fasting Blood biochemistry including total cholesterol (TC), low-density lipoprotein-cholesterol (LDL-C), high-density-lipoprotein cholesterol (HDL-C), triglycerides (TG)
Diabetes control | Change from baseline to 2 months
  Measured through glycated haemoglobin (%) in fasting state
Physical Activity | Change from baseline to 2 months
  Self-reported through the International Physical Activity Questionnaire, classifying the activity in three categories (low activity levels, moderate activity levels or high activity levels)
Physical Activity | Change from baseline to 2 months
  objectively assessed by accelerometer, to wear for seven consecutive days
Smoking Cessation | Change from baseline to 2 months
  Cigarette smoking habits quantified in pack-year and cigarettes per day, to measure exposure to tobacco
Depression and anxiety | Change from baseline to 2 months
  Psychosocial parameters assessed through the Hospital Anxiety and Depression Score questionnaire. Scores 0-14. A sub-scale score > 8 denotes anxiety or depression symptoms
Health Related Quality of Life | Change from baseline to 2 months
  Evaluated using the EuroQuol Five- Dimensional questionnaire ( EQ-5D-5L). It consists in five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ - Visual Analog Scale records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Fatigue | Change from baseline to 2 months
  Fatigue score evaluated by the specific item on the EORTC QLQ-C30 questionnaire (high score representing high level of symptomatology)
Health Literacy | Change from baseline to 2 months
  Assessed by the Newest Vital Sign questionnaire; range score 0-6 (high score corresponding to high health literacy)
Inflammatory markers- Interleukin-6 (IL-6) | Change from baseline to 2 months
  Blood samples collected to access plasma levels of IL-6
Inflammatory markers - High-sensitivity C-reactive protein | Change from baseline to 2 months
  Blood samples collected to access plasma levels of high-sensitivity C-reactive protein
Feasibility - Consent rate | Through study recruitment, up to 2 years
  number of patients who met inclusion criteria divided by the number who consented in writing to participate. Reasons for not participating in the study will be registered.
Testing and Intervention Adverse events | Change from baseline to 2 months
  all the events will be recorded and registered as "related" or "unrelated" to the intervention itself, as well as the impact for exercise concerns or other health intervention required
Feasibility - Retention rate | Change from baseline to 2 months
  number of participants who remained in the study (without formally drop out during intervention).
Feasibility - Intervention adherence | Change from baseline to 2 months
  total number of exercise sessions attended by participants allocated to this intervention group. Reasons for dropping out will be registered.
Feasibility - Completion rate | Change from baseline to 2 months
  number of patients that completed all the evaluations during the defined timeline.
Cost-effectiveness analysis | From baseline assessment up to 2 years
  Incremental cost per quality-adjusted life. Costs will be calculated from the provider perspective, which includes the costs incurred by the health institution providing health services; and from the societal perspective

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Vila Nova de Gaia Espinho, E.P.E., Vila Nova de Gaia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Viamonte SG, Joaquim AV, Alves AJ, Vilela E, Capela A, Ferreira C, Duarte BF, Rato ND, Teixeira MP, Tavares A, Santos M, Ribeiro F. Cardio-Oncology Rehabilitation for Cancer Survivors With High Cardiovascular Risk: A Randomized Clinical Trial. JAMA Cardiol. 2023 Dec 1;8(12):1119-1128. doi: 10.1001/jamacardio.2023.3558. PMID 37819656